CLINICAL TRIAL: NCT04234906
Title: Multicenter Study for the Prevention of Post-Operative Cardiac Arrhythmias
Brief Title: Prevention of Post-Operative Cardiac Arrhythmias
Acronym: POCA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeffrey Moak (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Moak, Director, Electrophysiology and Pacing, Principle Investigator, Clinical Professor, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013067
Record Dates: First submitted 2020-01-06; First posted 2020-01-21 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-12

CONDITIONS: Cardiac; Dysrhythmia, Postoperative; Congenital Heart Surgery
Keywords: Magnesium Sulfate; Dexedetomidine; anti-arrhythmic medications
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Dexmedetomidine; Magnesium Sulfate; Amiodarone; Procainamide

STUDY DESIGN:
Intervention Model Description: Two staged, prospective randomized clinical trial:
  Stage 1 targets prevention of post-operative arrhythmias.
  Stage 2 allows for re-randomization to secondary treatment for those subjects failing Stage 1, i.e. those patients that develop and require treatment of clinically significant post-operative cardiac arrhythmias with antiarrhythmic medication.
Masking Description: Patients will be randomized within each participating center, not by center, into study groups:
  Stage 1: Group 1 - Dexmedetomidine vs. Group 2- Magnesium Sulfate + Dexmedetomidine
  Stage 2: If clinically significant arrhythmias in need of treatment develop, patients will be randomized to Group 1 - amiodarone vs. procainamide.
  Randomization will occur through a module in Redcap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Stage 1, Group 1 - Dexmedetomidine (Active Comparator): Dexmedetomidine: 1 mcg/kg administered at end of cardiopulmonary bypass, followed by a 0.5 mcg/kg/h infusion for 72 h postoperatively or ready for extubation prior to 72 hour time period
  Interventions: Drug: Dexmedetomidine
- Stage 1, Group 2- Magnesium (Active Comparator): Magnesium Sulfate (50 mg/kg) bolus administered at the time of Aortic Cross Clamp Release, with continued administration for 72 hours postoperatively at a dose of 30 mg/kg/day.
  Interventions: Drug: Magnesium Sulfate
- Stage 2, AMIODARONE (Active Comparator): AMIODARONE I V Amiodarone 2.5 mg/kg administered over 30 minutes Second 2.5 mg/kg dose if needed over 30 minutes Continuous Intravenous Infusion 10-15 mg/kg/24 hours
  Interventions: Drug: Amiodarone
- Stage 2, PROCAINAMIDE (Active Comparator): PROCAINAMIDE IV Procainamide 10-15 mg/kg administered over 45 minutes Continuous Intravenous Infusion 20-50 mcg/kg/min
  Interventions: Drug: Procainamide

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine: 1 mcg/kg administered over 20 min peri-intubation period, followed by a 0.5 mcg/kg/h infusion for 72 h postoperatively or ready for extubation prior to 72 hour time period
  Other Names: Precedex
  Arms: Stage 1, Group 1 - Dexmedetomidine
Drug: Magnesium Sulfate — Magnesium Sulfate (50 mg/kg) bolus administered at the time of Aortic Cross Clamp Release, with continued administration for 72 hours postoperatively at a dose of 30 mg/kg/day
  Arms: Stage 1, Group 2- Magnesium
Drug: Amiodarone — I V Amiodarone 2.5 mg/kg administered over 30 minutes Second 2.5 mg/kg dose if needed over 30 minutes Continuous Intravenous Infusion 10-15 mg/kg/24 hours
  Arms: Stage 2, AMIODARONE
Drug: Procainamide — IV Procainamide 10-15 mg/kg administered over 45 minutes Continuous Intravenous Infusion 20-50 mcg/kg/min
  Other Names: Pronestyl
  Arms: Stage 2, PROCAINAMIDE

SUMMARY:
Aim 1: Primary Prevention of Post-operative Cardiac Arrhythmias

1. To evaluate the efficacy of dexmedetomidine vs. the combination of Magnesium Sulfate and dexmedetomidine for the prevention of post-operative cardiac arrhythmias in children and young adults undergoing open heart surgical repair for congenital or acquired heart disease using cardiopulmonary bypass. Dexmedetomidine is currently being administered to almost all patients after coming off cardiopulmonary bypass and in the CICU. For this aim, the investigator will be comparing dexmedetomidine administered alone or in combination with Magnesium Sulfate.
2. To evaluate medication safety based on the frequency of Serious Adverse Events (SAEs) and Adverse Events (AEs)

Aim 2: Secondary treatment of those Patients that develop a clinically significant arrhythmia despite having received either Dexmedetomidine alone or Magnesium Sulfate with Dexmedetomidine at the time of cardiac surgery

1. To evaluate the efficacy of intravenous (IV) Amiodarone vs. IV Procainamide for the control of postoperative cardiac arrhythmias developing after the failure of Stage 1, Preventative Trial. IV amiodarone and IV procainamide are standardly used treatment agents for the treatment of postoperative cardiac arrhythmias in this setting. The investigator will be assessing the comparative effectiveness of these agents in controlling post-operative cardiac arrhythmias.
2. To evaluate antiarrhythmic medication safety based on the frequency of SAEs and AEs

DETAILED DESCRIPTION:
Objective: Postoperative cardiac arrhythmias (POCA) are common in children undergoing congenital heart surgery using the heart-lung machine (cardiopulmonary bypass) and have been reported in 5-38% of patients. The occurrence of arrhythmias frequently delays the patient's postoperative recovery, prolongs Cardiac Intensive Care Unit (CICU) and hospital stay, increases costs for hospital care and increases postoperative morbidity and mortality.

Magnesium Sulfate has been one agent used to reduce the occurrence of postoperative arrhythmias. The investigators recently published a propensity-score matched study of the intra-operative administration of Magnesium Sulfate revealing that as many as one-third of pediatric patients at Children's National Hospital undergoing open-heart surgery using cardiopulmonary bypass have postoperative arrhythmias. The use of intraoperative Magnesium Sulfate was associated with a reduction in the occurrence of postoperative arrhythmias. However, despite the intraoperative use of Magnesium Sulfate there continued to be a fairly high residual occurrence rate of post-operative arrhythmias (total arrhythmia frequency -18%).

Dexmedetomidine has also been showed to reduce the occurrence of POCA and has become the preferred agent used for post-operative sedation and pain control. In several studies reported in the medical literature, dexmedetomidine has been found to decrease the occurrence of POCA, like Magnesium Sulfate.

In this IRB study, the investigator is proposing a clinical study to test if the investigator can further decrease the occurrence of postoperative arrhythmias. The investigator will be studying if Magnesium Sulfate administrated in conjunction with an intravenous anesthetic medication, known as dexmedetomidine, can further decrease the primary occurrence of post-operative arrhythmias. The investigator hypothesizes that the effect achieved with the simultaneous administration of Magnesium Sulfate and dexmedetomidine will be much greater than either medication used alone.

For those patients who fail preventative medical strategies and develop clinical significant post-operative arrhythmias in need of treatment, rescue arrhythmia treatment options include the use of potent anti-arrhythmic medications that can have very dramatic effects on the patient's heart rate and blood pressure (amiodarone or procainamide). Scant published data exists providing us with guidance on the comparative efficacy and safety of these agents in the postoperative cardiac surgical patient. The investigator will compare the efficacy and adverse effects of the two agents in treating clinically significant arrhythmias that occur despite trying to prevent their onset.

ELIGIBILITY:
Inclusion Criteria:

* 1) Any infant, child, adolescent, or young adult with congenital or acquired heart disease undergoing open heart surgical repair using cardiopulmonary bypass is eligible to be enrolled in this trial.
* 2) No age, gender or ethnic group restrictions.

Exclusion Criteria:

* 1) Non-cardiopulmonary bypass repair of a congenital or acquired cardiac defect.
* 2) Significant pre-operative arrhythmia history
* 3) Past history of adverse effect to any of the study medication agents

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 870 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Operative Cardiac Arrhythmias | 3 years
  The investigator will determine the incidence of cardiac arrhythmia in the two study groups (dexmedetomidine and magnesium sulfate). Statistical analysis will be performed to determine whether a statistical difference is detected between the two study groups. The occurrence of cardiac arrhythmias will be determined from continuous cardiac telemetry.

SECONDARY OUTCOMES:
Percent of Treatment Success Following IV Amiodarone or Procainamide Administration for Post-Operative Cardiac Arrhythmias. | 3 years
  The investigator will determine treatment success (as measured by the composite of complete or partial arrhythmia control) following the administration of either IV amiodarone or procainamide administration. Percent of treatment success will be determined by the composite success group divided by all given administered each anti-arrhythmic agent. Statistical analysis will be performed to determine whether a statistical difference is detected between the two study groups. Arrhythmia control will be determined from continuous cardiac telemetry.
Incidence of Adverse Effects following IV Amiodarone or Procainamide Administration | 3 years
  The investigator will determine the incidence of adverse effects (hypotension, bradycardia, or low cardiac output) following the administration of either IV amiodarone or procainamide. Statistical analysis will be performed to determine whether a statistical difference is detected between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Moak, Principal Investigator — Children's National Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rekawek J, Kansy A, Miszczak-Knecht M, Manowska M, Bieganowska K, Brzezinska-Paszke M, Szymaniak E, Turska-Kmiec A, Maruszewski P, Burczynski P, Kawalec W. Risk factors for cardiac arrhythmias in children with congenital heart disease after surgical intervention in the early postoperative period. J Thorac Cardiovasc Surg. 2007 Apr;133(4):900-4. doi: 10.1016/j.jtcvs.2006.12.011. PMID 17382623
- [Background] Hoffman TM, Bush DM, Wernovsky G, Cohen MI, Wieand TS, Gaynor JW, Spray TL, Rhodes LA. Postoperative junctional ectopic tachycardia in children: incidence, risk factors, and treatment. Ann Thorac Surg. 2002 Nov;74(5):1607-11. doi: 10.1016/s0003-4975(02)04014-6. PMID 12440616
- [Background] Dodge-Khatami A, Miller OI, Anderson RH, Goldman AP, Gil-Jaurena JM, Elliott MJ, Tsang VT, De Leval MR. Surgical substrates of postoperative junctional ectopic tachycardia in congenital heart defects. J Thorac Cardiovasc Surg. 2002 Apr;123(4):624-30. doi: 10.1067/mtc.2002.121046. PMID 11986588
- [Background] Cecchin F, Johnsrude CL, Perry JC, Friedman RA. Effect of age and surgical technique on symptomatic arrhythmias after the Fontan procedure. Am J Cardiol. 1995 Aug 15;76(5):386-91. doi: 10.1016/s0002-9149(99)80106-4. PMID 7639165
- [Background] Pfammatter JP, Wagner B, Berdat P, Bachmann DC, Pavlovic M, Pfenninger J, Carrel T. Procedural factors associated with early postoperative arrhythmias after repair of congenital heart defects. J Thorac Cardiovasc Surg. 2002 Feb;123(2):258-62. doi: 10.1067/mtc.2002.119701. PMID 11828284
- [Background] Moak JP, Arias P, Kaltman JR, Cheng Y, McCarter R, Hanumanthaiah S, Martin GR, Jonas RA. Postoperative junctional ectopic tachycardia: risk factors for occurrence in the modern surgical era. Pacing Clin Electrophysiol. 2013 Sep;36(9):1156-68. doi: 10.1111/pace.12163. Epub 2013 May 10. PMID 23662635
- [Background] He D, Aggarwal N, Zurakowski D, Jonas RA, Berul CI, Hanumanthaiah S, Moak JP. Lower risk of postoperative arrhythmias in congenital heart surgery following intraoperative administration of magnesium. J Thorac Cardiovasc Surg. 2018 Aug;156(2):763-770.e1. doi: 10.1016/j.jtcvs.2018.04.044. Epub 2018 Apr 18. PMID 29778339
- [Background] He D, Sznycer-Taub N, Cheng Y, McCarter R, Jonas RA, Hanumanthaiah S, Moak JP. Magnesium Lowers the Incidence of Postoperative Junctional Ectopic Tachycardia in Congenital Heart Surgical Patients: Is There a Relationship to Surgical Procedure Complexity? Pediatr Cardiol. 2015 Aug;36(6):1179-85. doi: 10.1007/s00246-015-1141-5. Epub 2015 Mar 12. PMID 25762470
- [Background] Lapsa J, Clark B, Chen YI, Moak JP. Incidence and risk factors for development of post-operative bradyarrhythmias following congenital and acquired cardiac disease repair in pediatric patients. Poster at APS, Baltimore, MD, 2019.
- [Background] El Amrousy DM, Elshmaa NS, El-Kashlan M, Hassan S, Elsanosy M, Hablas N, Elrifaey S, El-Feky W. Efficacy of Prophylactic Dexmedetomidine in Preventing Postoperative Junctional Ectopic Tachycardia After Pediatric Cardiac Surgery. J Am Heart Assoc. 2017 Mar 1;6(3):e004780. doi: 10.1161/JAHA.116.004780. PMID 28249845
- [Background] Chrysostomou C, Sanchez-de-Toledo J, Wearden P, Jooste EH, Lichtenstein SE, Callahan PM, Suresh T, O'Malley E, Shiderly D, Haney J, Yoshida M, Orr R, Munoz R, Morell VO. Perioperative use of dexmedetomidine is associated with decreased incidence of ventricular and supraventricular tachyarrhythmias after congenital cardiac operations. Ann Thorac Surg. 2011 Sep;92(3):964-72; discussion 972. doi: 10.1016/j.athoracsur.2011.04.099. PMID 21871284
- [Background] Chang PM, Silka MJ, Moromisato DY, Bar-Cohen Y. Amiodarone versus procainamide for the acute treatment of recurrent supraventricular tachycardia in pediatric patients. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):134-40. doi: 10.1161/CIRCEP.109.901629. Epub 2010 Mar 1. PMID 20194798
- [Background] Jian W, Su L, Yiwu L. The effects of magnesium prime solution on magnesium levels and potassium loss in open heart surgery. Anesth Analg. 2003 Jun;96(6):1617-1620. doi: 10.1213/01.ANE.0000065444.21593.23. PMID 12760983
- [Background] Manrique AM, Arroyo M, Lin Y, El Khoudary SR, Colvin E, Lichtenstein S, Chrysostomou C, Orr R, Jooste E, Davis P, Wearden P, Morell V, Munoz R. Magnesium supplementation during cardiopulmonary bypass to prevent junctional ectopic tachycardia after pediatric cardiac surgery: a randomized controlled study. J Thorac Cardiovasc Surg. 2010 Jan;139(1):162-169.e2. doi: 10.1016/j.jtcvs.2009.07.064. Epub 2009 Oct 12. PMID 19819469
- [Background] Dittrich S, Germanakis J, Dahnert I, Stiller B, Dittrich H, Vogel M, Lange PE. Randomised trial on the influence of continuous magnesium infusion on arrhythmias following cardiopulmonary bypass surgery for congenital heart disease. Intensive Care Med. 2003 Jul;29(7):1141-4. doi: 10.1007/s00134-003-1802-3. Epub 2003 May 28. PMID 12774159
- [Background] Lee HY, Ghimire S, Kim EY. Magnesium supplementation reduces postoperative arrhythmias after cardiopulmonary bypass in pediatrics: a metaanalysis of randomized controlled trials. Pediatr Cardiol. 2013 Aug;34(6):1396-403. doi: 10.1007/s00246-013-0658-8. Epub 2013 Feb 27. PMID 23443885
- [Background] Dorman BH, Sade RM, Burnette JS, Wiles HB, Pinosky ML, Reeves ST, Bond BR, Spinale FG. Magnesium supplementation in the prevention of arrhythmias in pediatric patients undergoing surgery for congenital heart defects. Am Heart J. 2000 Mar;139(3):522-8. doi: 10.1016/s0002-8703(00)90097-8. PMID 10689268
- [Background] Verma YS, Chauhan S, Gharde P, Lakshmy R, Kiran U. Role of magnesium in the prevention of postoperative arrhythmias in neonates and infants undergoing arterial switch operation. Interact Cardiovasc Thorac Surg. 2010 Nov;11(5):573-6. doi: 10.1510/icvts.2010.239830. Epub 2010 Aug 5. PMID 20688775
- [Background] Fairley JL, Zhang L, Glassford NJ, Bellomo R. Magnesium status and magnesium therapy in cardiac surgery: A systematic review and meta-analysis focusing on arrhythmia prevention. J Crit Care. 2017 Dec;42:69-77. doi: 10.1016/j.jcrc.2017.05.038. Epub 2017 Jun 21. PMID 28688240
- [Background] Li X, Zhang C, Dai D, Liu H, Ge S. Efficacy of dexmedetomidine in prevention of junctional ectopic tachycardia and acute kidney injury after pediatric cardiac surgery: A meta-analysis. Congenit Heart Dis. 2018 Sep;13(5):799-807. doi: 10.1111/chd.12674. Epub 2018 Sep 27. PMID 30260073
- [Background] Gautam NK, Turiy Y, Srinivasan C. Preincision Initiation of Dexmedetomidine Maximally Reduces the Risk of Junctional Ectopic Tachycardia in Children Undergoing Ventricular Septal Defect Repairs. J Cardiothorac Vasc Anesth. 2017 Dec;31(6):1960-1965. doi: 10.1053/j.jvca.2017.04.010. Epub 2017 Apr 10. PMID 28774644
- [Background] Mahmoud AB, Tantawy AE, Kouatli AA, Baslaim GM. Propranolol: a new indication for an old drug in preventing postoperative junctional ectopic tachycardia after surgical repair of tetralogy of Fallot. Interact Cardiovasc Thorac Surg. 2008 Apr;7(2):184-7. doi: 10.1510/icvts.2007.160945. Epub 2007 Dec 18. PMID 18089616
- [Background] Shuplock JM, Smith AH, Owen J, Van Driest SL, Marshall M, Saville B, Xu M, Radbill AE, Fish FA, Kannankeril PJ. Association between perioperative dexmedetomidine and arrhythmias after surgery for congenital heart disease. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):643-50. doi: 10.1161/CIRCEP.114.002301. Epub 2015 Apr 15. PMID 25878324
- [Background] Amrousy DE, Elshehaby W, Feky WE, Elshmaa NS. Safety and Efficacy of Prophylactic Amiodarone in Preventing Early Junctional Ectopic Tachycardia (JET) in Children After Cardiac Surgery and Determination of Its Risk Factor. Pediatr Cardiol. 2016 Apr;37(4):734-9. doi: 10.1007/s00246-016-1343-5. Epub 2016 Jan 27. PMID 26818850
- [Background] Lakatos E. Sample sizes based on the log-rank statistic in complex clinical trials. Biometrics. 1988 Mar;44(1):229-41. PMID 3358991
- [Background] Lakatos E. Designing complex group sequential survival trials. Stat Med. 2002 Jul 30;21(14):1969-89. doi: 10.1002/sim.1193. PMID 12111882